CLINICAL TRIAL: NCT00504452
Title: An Open-Label, Multicenter, Mechanism Validation Study to Evaluate the Safety, Efficacy and Tolerability of KP-1461 as Monotherapy for 124 Days in Antiretroviral-experienced, HIV-1-infected Subjects
Brief Title: Safety and Efficacy Study of KP-1461 to Treat ART-Experienced HIV+ Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Corroboration of supporting in vitro data
  - Data successfully corroborated 2009
Sponsor: Koronis Pharmaceuticals. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KP-1461-201
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2008-11

CONDITIONS: HIV Infections
Keywords: HIV; viral; Viral decay acceleration; ART; HAART; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — KP 1461

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: KP-1461 — Oral dosage, 1600 mg bid for 124 days

SUMMARY:
The primary purpose of the study is to investigate the safety and efficacy of KP-1461 given every 12 hours for 124 days to HIV+ patients who have failed multiple antiretroviral regimens.

DETAILED DESCRIPTION:
KP-1461 is a prodrug of KP-1212 triphosphate, a unique nucleoside that is incorporated into the HIV viral genome resulting in an accumulation of nucleic substitutions that interfere with viral replication. The study is designed to investigate the safety and antiviral activity for 124 days in antiretroviral-experienced HIV-1-infected subjects. By inducing additional mutagenic events in the viral genome, viral decay accelerators such as KP-1212 may force the virus to exceed the threshold of nonviability.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic HIV-1-infected individuals who are treatment-experienced and who have not been on ART for at least 16 weeks.
* Have documented prior non-suppressive ART including at least 1 NRTI, 1 NNRTI and 2 PIs; or have documented prior ART resistance to at least 1 NRTI, 1 NNRTI and 1 PI; AND in the opinion of the investigator, have few, if any, effective treatment options available.
* Have >2,500 copies/mL of HIV-1 RNA at screening.
* Have a stable CD4 cell count while off ART and >250 cells/mL at screening.
* Have no clinically significant findings on screening evaluations.

Exclusion Criteria:

* Have a current or recent opportunistic infection that, in the opinion of the investigator, is not being controlled by medication.
* Have any condition that, in the opinion of the investigator, could compromise subject safety or adherence to the protocol.
* Have a documented positive test for hepatitis B surface antigen, or have received any antiviral therapy for hepatitis C <6 weeks prior to study drug administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-07; Primary Completion 2008-09 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of KP-1461 for 124 days in treatment-experienced, HIV-1-infected subjects. | 124 days

SECONDARY OUTCOMES:
To evaluate the antiviral activity (eg., CD4 count, HIV RNA count) of KP-1461 for 124 days in treatment-experienced, HIV-1-infected subjects. | 124 days

CONTACTS AND LOCATIONS:
Locations (31):
- United States (30):
  - Health for Life Clinic, Little Rock, Arkansas
  - Living Hope Clinical Foundation, Long Beach, California
  - Light Source Medical/U. of Southern California, Los Angeles, California
  - ACTU at CARES/UC Davis, Sacramento, California
  - UCSD Antiviral Research Center, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - Dupont Circle Physician's Group, Washington D.C., District of Columbia
  - Whitman-Walker Clinic, Washington D.C., District of Columbia
  - Comprehensive Care Center -- HIV Clinical Research, Fort Lauderdale, Florida
  - Wohlfeiler, Piperato and Associates, LLC, North Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Treasure Coast Infectious Disease Consultants, Vero Beach, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Northstar Medical Center, Chicago, Illinois
  - University of Kansas School of Medicine - PriVia, The Research Centers of Via Christi, Wichita, Kansas
  - Institute of Human Virology, University of Maryland, Baltimore, Maryland
  - Community Research Initiative of New England, Boston, Massachusetts
  - Dybedal Center for Clinical Research, Kansas City University of Medicine and Biosciences, Kansas City, Missouri
  - St. Michael's Medical Center, Newark, New Jersey
  - Southwest CARE Center, Santa Fe, New Mexico
  - Albany Medical College, Albany, New York
  - AIDS Community Research Initiative of America, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Thomas Jefferson University, Division of Infectious Disease, Philadelphia, Pennsylvania
  - Charlton Methodist Hospital, Dallas, Texas
  - University of Texas Health Science Center, Houston, Texas
  - CARE-ID, Annandale, Virginia
  - University of Washington AIDS Clinical Trials Unit, Seattle, Washington
- Clinical Research Puerto Rico, Inc., San Juan, Puerto Rico

REFERENCES:
- See also: Results on drug activity in patients who completed treatment — http://www.plosone.org/article/info%3Adoi%2F10.1371%2Fjournal.pone.0015135